CLINICAL TRIAL: NCT05409482
Title: A Real-world Study of Camrelizumab Combined With Apatinib Mesylate in Unresectable Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other)
Collaborators: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongyi Zeng, director, Meng Chao Hepatobiliary Hospital of Fujian Medical University
Other Study IDs: 22-OBU-FJ-CA-ALL-001
Record Dates: First submitted 2022-05-25; First posted 2022-06-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the efficacy and safety of camrelizumab combined with apatinib mesylate in the treatment of unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
Combination therapy for patients with unresectable liver cancer is the future trend, and with the development of therapeutic drugs for liver cancer, especially molecular targeted drugs and immunotherapy drugs, the effective rate of liver cancer treatment has been significantly improved, and the treatment of unresectable liver cancer has gradually changed. possible. Therefore, for patients with unresectable liver cancer, how to choose a combined treatment plan will be an important means to improve the therapeutic effect of liver cancer, and it is also a hot spot in the field of clinical research on liver cancer in recent years.

Based on the above research background, this study is now designed as a non-intervention, selecting patients with unresectable hepatocellular carcinoma as the research subjects to analyze the efficacy and safety of camrelizumab combined with apatinib mesylate. In order to bring more long-term benefits to patients with unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years old ≤ age ≤ 75 years old, both male and female;
2. Strictly meet the clinical diagnostic criteria of the "Guidelines for the Diagnosis and Treatment of Primary Liver Cancer" (2022 Edition) or hepatocellular carcinoma patients diagnosed by histopathological or cytological examinations , and at least one measurable lesion (according to the mRECIST1.1 standard, the long diameter of the measurable lesion on spiral CT scan is ≥10mm or the short diameter of the malignant lymph node is ≥15mm);
3. Not previously accepted Patients with hepatocellular carcinoma who have progressed/intolerable and unresectable after systemic therapy or first-line systemic therapy;
4. CNLC stage IIb-IIIb;
5. Child-Pugh liver function grade A or B (5- 7 points);
6. ECOG PS score 0-1 points;
7. Expected survival period ≥ 12 weeks;
8. If the patient has active hepatitis B virus (HBV) infection: if HBV-DNA ≤ 2000, you can start directly Treatment; if HBV-DNA>2000, antiviral treatment should be given for one week before starting treatment;
9. The subjects volunteered to join the study, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. Patients with contraindications to immunotherapy, including but not limited to the following: post-transplantation patients, patients with severe autoimmune diseases, patients with organ failure, patients who have previously experienced adverse reactions of grade 4 or above using immunotherapy, and uncontrolled infectious diseases;
3. Use immunosuppressive or systemic hormone therapy within 14 days before enrollment to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other equivalent hormones);
4. It has been confirmed that camrelizumab Patients who are allergic to injections, apatinib mesylate tablets and their excipients, or are allergic to other monoclonal antibodies;
5. Patients with impaired consciousness or inability to cooperate with treatment, combined with mental illness;
6. Patients who have participated in other clinical trials in the past three months;
7. Severe liver, kidney, heart, lung, brain and other major organ failure;
8. According to the investigator's judgment, patients with other serious concomitant diseases that endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（PFS） | Up to 2 years
  PFS was defined as the subject's date from the date of the first dose to the date of the first documented tumor progression (as assessed by mRECIST criteria, with or without continuation of treatment) or the date of death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Objective response rate（ORR） | Up to 2 years
  Refers to the proportion of all subjects with the best overall response (BOR) as complete remission (CR) or partial remission (PR) according to mRECIST 1.1 criteria.
Disease control rate（DCR） | Up to 2 years
  Refers to the proportion of all subjects with the best overall response (BOR) according to mRECIST criteria as complete remission (CR), partial remission (PR) and stable disease (SD).
Overall survival（OS） | Up to 8 years
  Defined as the time from the date of the first dose to the death of the subject from any cause.
Occurence of AE and SAE | Up to 2 years
  Occurence of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）

CONTACTS AND LOCATIONS:
Overall Officials: Wu h Guo, Study Director — Mengchao Hepatobiliary Hospital, Fujian Medical University; Zhi bo Zhang, Study Director — First Affiliated Hospital of Fujian Medical University; Yi p Chen, Study Director — First Affiliated Hospital of Fujian Medical University; Ning Huang, Study Director — Union Hospital, Affiliated to Fujian Medical University; Mao l Yan, Study Director — Fujian Provincial Hospital; Zhu t Fang, Study Director — Fujian Provincial Hospital; Hui Zhang, Study Director — Fujian Cancer Hospital; Xiao j Zhang, Study Director — The 900th Hospital of the Joint Logistics Support Force; Ling q Yan, Study Director — Fuqing City Hospital; Yan m Zhou, Study Director — The First Affiliated Hospital of Xiamen University; Yong yi Zeng, Principal Investigator — Mengchao Hepatobiliary Hospital, Fujian Medical University; Ping g Liu, Study Director — Zhongshan Hospital Affiliated to Xiamen University; Fu q Wang, Study Chair — Xiamen Hospital of Traditional Chinese Medicine; Bo h Zhang, Study Director — Zhongshan Hospital (Xiamen), Fudan University; Cong r Wang, Study Director — Quanzhou First Hospital; Wei Wang, Study Director — The Second Affiliated Hospital of Fujian Medical University; Yu f Chen, Study Director — Zhangzhou Hospital; Shao w Zhuang, Study Chair — Zhangzhou Hospital; Jian f Zhao, Study Director — Affiliated Hospital of Putian University; Jia f Chen, Study Director — Putian First Hospital; Wen l Zeng, Study Director — Longyan Second Hospital; Yong z Wang, Study Director — Sanming Second Hospital; Wen f Wu, Study Director — Nanping Second Hospital; Wen x Xie, Study Director — Fuding City Hospital; Feng Lin, Study Director — Ningde Mindong Hospital
Locations (1):
- Mengchao Hepatobiliary Hospital, Fujian Medical University, Fuzhou, Fujian, China